CLINICAL TRIAL: NCT03035513
Title: Diffusion Tensor Imaging of the Thalamo-cortical Network in Epilepsy With Continuous Spikes and Waves During Sleep
Brief Title: Diffusion Tensor Imaging in Epilepsy With Continuous Spikes and Waves During Sleep
Acronym: POCS-DTI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0299; 2016-A01149-42 (Other: 2016-A01149-42)
Record Dates: First submitted 2017-01-13; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Cryptogenic Epilepsy
Keywords: Continuous spikes; Epilepsy; Nervous system disease; Neuronal plasticity; Diffusion MRI; Functional MRI; waves during slow sleep (CSWS)
MeSH Terms: conditions — Epilepsy; Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- CSWS patients: The data of CSWS patients will be statistically compared to healthy volunteers
  Interventions: Other: Continuous spikes and waves during slow sleep (CSWS)
- healthy volunteers: The data of CSWS patients will be statistically compared to healthy volunteers
  Interventions: Other: Continuous spikes and waves during slow sleep (CSWS)

INTERVENTIONS:
Other: Continuous spikes and waves during slow sleep (CSWS)

SUMMARY:
Continuous Spikes and Waves during Sleep (CSWS) is a rare paediatric epileptic encephalopathy. Even if the correlation between the severity of the epilepsy and the cognitive consequences is well established, the mechanisms involved in epileptic cognitive degradation are complex and poorly understood. In CSWS, there are many arguments for the implication of cortical and subcortical cerebral structures. Among them the thalamus seems to play a crucial role. In fact it is strongly implicated in the sleep and this function is determining for learning. Moreover, it is part of the propagation pathway of generalized forms of epilepsy like absences in animal studies. Unfortunately there is no animal model for CSWS to confirm this theory. In human studies, few cases are caused by thalamic injuries but most of the time conventional MRI is normal. Despite few literature on CSWS, some studies reported abnormal functional connectivity especially in the thalamus.

The investigators hypothesize that the first utilisation of diffusion tensor imaging (DTI) and tractography will be useful in CSWS to confirm the implication of a cortico-thalamo-cortical network showing an abnormal structural connectivity. The investigators will try to determinate if a particular thalamic nucleus is concerned and demonstrate a link between the disease severity (duration and cognitive consequences) and the importance of structural abnormalities.

Using resting state functional MRI (fMRI), the investigators will also try to investigate the default mode network. Its implication was also suggested in the literature.

DETAILED DESCRIPTION:
Continuous Spikes and Waves during Sleep (CSWS) is a rare paediatric epileptic encephalopathy. Even if the correlation between the severity of the epilepsy and the cognitive consequences is well established, the mechanisms involved in epileptic cognitive degradation are complex and poorly understood. In CSWS, there are many arguments for the implication of cortical and subcortical cerebral structures. Among them the thalamus seems to play a crucial role. In fact it is strongly implicated in the sleep and this function is determining for learning. Moreover, it is part of the propagation pathway of generalized forms of epilepsy like absences in animal studies. Unfortunately there is no animal model for CSWS to confirm this theory. In human studies, few cases are caused by thalamic injuries but most of the time conventional MRI is normal. Despite few literature on CSWS, some studies reported abnormal functional connectivity especially in the thalamus.

The investigators hypothesize that the first utilisation of diffusion tensor imaging (DTI) and tractography will be useful in CSWS to confirm the implication of a cortico-thalamo-cortical network showing an abnormal structural connectivity. The investigators will try to determinate if a particular thalamic nucleus is concerned and demonstrate a link between the disease severity (duration and cognitive consequences) and the importance of structural abnormalities.

Using resting state functional MRI (fMRI), the investigators will also try to investigate the default mode network. Its implication was also suggested in the literature.

ELIGIBILITY:
Inclusion Criteria:

* - for the patients, diagnosis of CSWS according to the current diagnostic criteria (ILAE 2001)
* minimal age of 5 years old
* written consent to participate in the study from the subjects who could write and/or from the parents or legal representative

Exclusion Criteria:

* rejection of the patient or its legal representative
* no respect of inclusion criteria

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients, diagnosis of CSWS according to the current diagnostic criteria (ILAE 2001)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Structural connectivity of the thalamo-cortical network | at day 1
  Structural connectivity of the thalamo-cortical network will be assessed using DTI fractional anisotropy.
  The data of CSWS patients will be statistically compared to healthy volunteers

SECONDARY OUTCOMES:
Some comparisons with electrophysiological and neuropsychological data will be done | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Dominique ROSENBERG, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France